CLINICAL TRIAL: NCT06728670
Title: Pharmacokinetic Study and Clinical Efficacy Observation of Different Routes of Tranexamic Acid Infusion in Advanced Ovarian Cancer Cell Reduction Surgery
Brief Title: Pharmacokinetic Study of Tranexamic Acid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Zhu Yejing, MD, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB-2024-1034
Record Dates: First submitted 2024-11-23; First posted 2024-12-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Neoplasm Epithelial
Keywords: Tranexamic acid; pharmacokinetics

STUDY DESIGN:
Intervention Model Description: Intravenous TXA injection group and intramuscular TXA injection group.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous infusion of TXA (Active Comparator): Slowly infuse 1g TXA at a rate of approximately 1 ml/min.
  Interventions: Behavioral: Tranexamic acid Intravenous Infusion
- Intramuscular injection of TXA (Experimental): 1g TXA is administered with twice intramuscular injections, and each injection takes no more than 30 seconds. The injection site is chosen as the deltoid or lateral thigh muscle.
  Interventions: Behavioral: TXA intramuscular injection

INTERVENTIONS:
Behavioral: Tranexamic acid Intravenous Infusion — A slow intravenous infusion of 1g TXA was administered at a rate of about 1ml/min.
  Arms: Intravenous infusion of TXA
Behavioral: TXA intramuscular injection — 5ml intramuscular injections of TXA with twice, each injection time no more than 30 seconds, the injection site was selected as triangle
  Arms: Intramuscular injection of TXA

SUMMARY:
Tranexamic acid is an effective anti fibrinolytic drug. Clinical studies have found that intravenous injection of tranexamic acid is more effective in reducing blood loss and transfusion in patients with advanced ovarian cancer, without increasing the risk of postoperative complications. Different surgeries and administration routes have an impact on the pharmacokinetics and pharmacodynamics of TXA. At present, there is little data on the pharmacokinetics of intramuscular injection of TXA, and almost all of the data comes from males. For ovarian cancer patients, there are currently no reports on the pharmacokinetics of TXA through different routes of administration, such as intramuscular and intravenous administration. Therefore, the investigators chose ovarian cancer patients and administered it through different routes of intravenous and intramuscular injection.

DETAILED DESCRIPTION:
The investigators plan to recuit 30 patients, administered TXA through different routes of administration. Then Pharmacokinetic parameters of different TXA administration routes were recorded. To study the effects of different TXA administration routes on intraoperative blood loss, transfusion volume and postoperative adverse outcomes (thrombosis, etc.) in ovarian cancer patients undergoing cell reduction surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult women aged 20-64 diagnosed with advanced ovarian cancer undergoing cytoreductive surgery
2. The cancer stage is III-IV
3. ASA classification II-III
4. Surgical duration>2 hours

Exclusion Criteria:

1. Renal dysfunction (serum creatinine>200 mmol/L) or liver dysfunction (Child Turcote classification>6)
2. Has a history of serious mental illness or disorders, epilepsy, visual impairment
3. Previous or current bleeding disorders, coagulation dysfunction, or thromboembolic events
4. Lower limb venous thrombosis
5. Anticoagulants or antifibrinolytic drugs used before surgery within the past month
6. Allergic to TXA

Ages: 20 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Elimination clearance rate (CL) of tranexamic acid | Before administration, 15minutes after administration, 45minutes after administration, 90minutes after administration, 3hours after administration, 6hours after administration and 24hours after administration
  Patients were enrolled and screened during preoperative anaesthesia visit. The enrolled patients were randomly divided into IV TXA injection group and intramuscular TXA injection group. All blood samples were centrifuged and preserved for later testing,Nonlinear mixed-effects pharmacokinetic modeling was performed on the compartmental population pharmacokinetic data using the Monolix 2020R1 program.
Interventricular clearance rate (Q) of tranexamic acid | Before administration, 15minutes after administration, 45minutes after administration, 90minutes after administration, 3hours after administration, 6hours after administration and 24hours after administration
  Patients were enrolled and screened during preoperative anaesthesia visit. The enrolled patients were randomly divided into IV TXA injection group and intramuscular TXA injection group. All blood samples were centrifuged and preserved for later testing,Nonlinear mixed-effects pharmacokinetic modeling was performed on the compartmental population pharmacokinetic data using the Monolix 2020R1 program.
Central ventricular volume (Vc) of tranexamic acid | Before administration, 15minutes after administration, 45minutes after administration, 90minutes after administration, 3hours after administration, 6hours after administration and 24hours after administration
  Patients were enrolled and screened during preoperative anaesthesia visit. The enrolled patients were randomly divided into IV TXA injection group and intramuscular TXA injection group. All blood samples were centrifuged and preserved for later testing,Nonlinear mixed-effects pharmacokinetic modeling was performed on the compartmental population pharmacokinetic data using the Monolix 2020R1 program.
peripheral ventricular volume (Vp) of tranexamic acid | Before administration, 15minutes after administration, 45minutes after administration, 90minutes after administration, 3hours after administration, 6hours after administration and 24hours after administration
  Patients were enrolled and screened during preoperative anaesthesia visit. The enrolled patients were randomly divided into IV TXA injection group and intramuscular TXA injection group. All blood samples were centrifuged and preserved for later testing,Nonlinear mixed-effects pharmacokinetic modeling was performed on the compartmental population pharmacokinetic data using the Monolix 2020R1 program.

SECONDARY OUTCOMES:
Intraoperative blood loss | during operative period
  blood should be taken before surgery for Hb or Hct measurements to determine the patient's current blood dilution or concentration.The calculation formula: estimated blood loss (ml) = (preoperative or estimated Hct - measured Hct) / preoperative or estimated Hctx weight (kg) x 7% x 1000.
Blood transfusion volume | during operative period
  The total volume of blood transfused during the operation was calculated, encompassing red blood cells, plasma, and cryoprecipitate.

OTHER OUTCOMES:
New postoperative thrombotic complications | within 30 days after surgery.
  ncidence of complications (new thrombus) are detected by vascular ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Result] Vergote I, Coens C, Nankivell M, Kristensen GB, Parmar MKB, Ehlen T, Jayson GC, Johnson N, Swart AM, Verheijen R, McCluggage WG, Perren T, Panici PB, Kenter G, Casado A, Mendiola C, Stuart G, Reed NS, Kehoe S; EORTC; MRC CHORUS study investigators. Neoadjuvant chemotherapy versus debulking surgery in advanced tubo-ovarian cancers: pooled analysis of individual patient data from the EORTC 55971 and CHORUS trials. Lancet Oncol. 2018 Dec;19(12):1680-1687. doi: 10.1016/S1470-2045(18)30566-7. Epub 2018 Nov 6. PMID 30413383